CLINICAL TRIAL: NCT04003428
Title: Perioperative Evaluation of High Intensity Focalized Ultrasound for Adjuvant Management of Placenta Accreta: a Clinical Feasibility Study
Brief Title: Feasibility of HIFU for Management of Placenta Accreta (HIFU-ACCRETA)
Acronym: HIFU-ACCRETA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lapsed Authorization (no patient)
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0335; 2017-A01376-47 (Other: ANSM)
Record Dates: First submitted 2019-04-25; First posted 2019-07-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Placenta Accreta
Keywords: High Intensity Focused Ultrasound (HIFU); Placenta accreta; Feasibility; Safety
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Per-caesarean HIFU shots (Experimental): Adjuvant treatment with High Intensity Focused Ultrasound (HIFU) performed the day of the scheduled childbirth, after confirmation of placenta accreta, and after fetal extraction by caesarian section.
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — HIFU shots will be performed on the placental tissue to produce necrotic lesions of approximately 30% of the total volume. A latency time of 2 minutes between each shot will be observed to avoid the accumulative heat effect, and to ensure optimal positioning of the treatment probe. The maximum duration of the operating time for HIFU shooting shall not exceed 60 minutes.

SUMMARY:
Placental accretion during pregnancy refers to an abnormally deep insertion of the placenta into the uterus, leading to the impossibility of removing the placenta without inducting uterine or surrounding organs lesions. The management of these patients is complex, with two options during caesarean section: hysterectomy or uterine conservative surgery in which the placenta is let in the uterine cavity. These are both at risk of complications, including severe hemorrhage.

High Intensity Focused Ultrasound (HIFU) principle is based on the focusing of ultrasonic waves in a focal zone causing a rapid rise in temperature in the targeted area. This focus results in the creation of a coagulation necrosis tissue lesion. This procedure is guided in real time by an integrated ultrasound imaging cell.

The investigators hypothesized that HIFU shots would accelerate the process of placental involution when the placenta is let in the uterine cavity, increasing the chances of uterine preservation and reducing the infectious and hemorrhagic risks in the short and medium term. The aim of this study is to confirm the feasibility and safety of the use of HIFU as a per-caesarean adjuvant treatment for management of placenta accrete let in the uterus for a conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman aged 18 years or older, with a suspicion of placental accretion observed with usual imaging tests (ultrasound, MRI)
* Single pregnancy (singleton)
* For whom a caesarean section has been scheduled
* Wishing to try to preserve her uterus
* Affiliated to a social security scheme or similar
* Having signed informed consent for participation in the study

Exclusion Criteria:

* Major patient protected by law, under guardianship or curatorship
* Patient participating in other interventional research that may interfere with this research
* Placental tumor identified in antenatal
* Grade 3 placental calcification
* Presence of a catheter, stent or vascular prosthesis close to the uterus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Success of HIFU per-caesarean shots | Up to 30 days after procedure
  Number of patients for whom: the probe is positioned in contact with the uterine serosa; and, one or more lesions of at least 1 cm each are visible on intraoperative ultrasound; and, total intervention time is 60 minutes maximum; and, no lesion are visible on the uterus; and, constants are maintained during the intervention; and, no related complication occurred during the intervention.

SECONDARY OUTCOMES:
Ultrasound characteristics of placental lesions produced over time | Up to 6 months after procedure
MRI characteristics of placental lesions produced over time | Up to 6 months after procedure
Characteristics of lesions produced by macroscopic and microscopic pathological examination of the placenta (only in case of hysterectomy) | Up to 6 months after procedure
Spontaneous uterine vacuity | Up to 6 months after procedure
  evaluated by endovaginal ultrasound examination. This examination will be supplemented by a liquid contrast ultrasound in accordance with standard clinical practices to identify the possible presence of synechia
Spontaneous uterine vacuity delay | Up to 6 months after procedure
  measured in daytime. This is an estimate. After surgery on the uterus (e.g. hysterectomy, hysteroscopy, aspiration-curetage endo-uterin) it is considered that spontaneous uterine emptiness is not obtained.
Occurrence of a complication (hemorrhage, infection or other) | Up to 6 months after procedure